CLINICAL TRIAL: NCT01592318
Title: An Up to Two-Part Relative Bioavailability Study of Ritonavir-Boosted Danoprevir Fixed Dose Combination Tablets as Compared to the Reference Phase 2 Ad Hoc Combination Tablets in Healthy Adult Volunteers
Brief Title: A Study of The Relative Bioavailability of Ritonavir-Boosted Danoprevir Fixed Dose Combination Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28136
Record Dates: First submitted 2012-04-24; First posted 2012-05-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ritonavir

ARMS (2):
- DNV + r reference (Active Comparator)
  Interventions: Drug: danoprevir; Drug: ritonavir
- DNV/r fixed dose combination (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — Fixed dose combination tablet with ritonavir, single oral dose
  Arms: DNV/r fixed dose combination
Drug: danoprevir — Reference tablet, single oral dose
  Arms: DNV + r reference
Drug: ritonavir — Fixed dose combination tablet with danoprevir, single oral dose
  Arms: DNV/r fixed dose combination
Drug: ritonavir — Reference tablet, single oral dose
  Arms: DNV + r reference

SUMMARY:
This randomized, open-label, crossover study will evaluate the relative bioavailability of ritonavir-boosted danoprevir fixed dose combination tablets (FDC) as compared to ad hoc combination of reference tablets of danoprevir and ritonavir in healthy volunteers. Subjects will be randomized to 1 of 6 treatment sequences to receive single oral doses of either an FDC of danoprevir and ritonavir or danoprevir and ritonavir as separate tablets. In a crossover design, subjects will participate in 3 study periods with at least a 7-day washout between periods. In Part 2, single dose administration of film-coated FDCs will be compared to reference tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers, 18 to 55 years of age
* Body weight >/= 50.0 kg
* Body mass index (BMI) 18.0 - 32.0 kg/m2
* Healthy non-smoking subjects. Healthy status will be defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history and a complete physical examination
* Medical history without major, recent, or ongoing pathology
* Females of childbearing potential and males and their female partners of childbearing potential must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last drug administration

Exclusion Criteria:

* Pregnant or lactating women or males with female partners who are pregnant or lactating
* Any history of clinically significant cardiovascular or cerebrovascular disease, hypertension, and/or infections
* Positive result for drugs of abuse at screening or prior to admission to the clinical site during any study period
* Positive for hepatitis B, hepatitis C or HIV infection
* Current smokers or subjects who have discontinued smoking less than 6 months prior to first dose of study medication
* Use of hormonal contraceptives (e.g. birth control pills, patches, injectable, implantable devices) within 30 days before the first dose of study medication
* Use of an investigational drug or device within 30 days of the first dose of study medication (6 months for biologic therapies) or 5 half-lives of the investigational drug, whichever is longer
* History of drug-related allergic reactions or hepatotoxicity
* History (within 3 months of screening) of alcohol consumption exceeding 2 standard drinks per day on average

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of danoprevir: Area under the concentration-time curve (AUC) | Pre-dose and up to 24 hours post-dose Days 1, 8 and 15
Pharmacokinetics of ritonavir: Area under the concentration-time curve (AUC) | Pre-dose and up to 24 hours post-dose Days 1, 8 and 15

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand